CLINICAL TRIAL: NCT01417663
Title: Combining Exercise Training With a Drug to Break AGE-crosslinks; Effects on Cardiovascular Structure and Function and Related Mechanisms
Brief Title: Effects of Exercise Training and AGE-crosslink Breaker on Cardiovascular Structure and Function
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Heart Foundation (Other); Synvista Therapeutics, Inc (Industry)
Responsible Party: Principal Investigator, Maria Hopman, Prof.Dr. M.T.E. Hopman, Radboud University Medical Center
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ALT-711-0529B
Record Dates: First submitted 2011-06-17; First posted 2011-08-16 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-09

CONDITIONS: Cardiovascular Disease; Aging; Endothelial Dysfunction; Physical Activity
Keywords: Aging; Cardiovascular disease; Endothelial function; Physical activity; Advanced Glycation Endproducts; AGE crosslink breakers
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity | interventions — alagebrium; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alagebrium (Placebo Comparator): In this study there will be four different groups:
  One Alagebrium 100 mg twice daily and exercise training 3x/week Two Placebo twice daily and exercise training 3x/week Three Alagebrium 100 mg twice daily and no exercise training Four Placebo twice daily and no exercise training
  Interventions: Drug: Alt-711; Behavioral: Physical exercise training
- Exercise training (Other): In this study there will be four different groups:
  One Alagebrium 100 mg twice daily and exercise training 3x/week Two Placebo twice daily and exercise training 3x/week Three Alagebrium 100 mg twice daily and no exercise training Four Placebo twice daily and no exercise training
  Interventions: Drug: Alt-711; Behavioral: Physical exercise training

INTERVENTIONS:
Drug: Alt-711 — Alt-711, also known as Alagebrium, an AGE-crosslink breaker, will be given twice daily 100mg
  Other Names: AGE crosslink breaker; Alagebrium; 4,5-dimethyl-3-(2-oxo-2-phenylethyl)-thiazolium chloride
Behavioral: Physical exercise training — Exercise training will be given three times a week for 45 minutes per training session. The heart rate reserve will be slowly increased from 70% to 85%.
  Other Names: Exercise training; Cardiopulmonary fitness training; Cycloergometer

SUMMARY:
Healthy but sedentary aging leads to increased morbidity and mortality of cardiovascular disease. This is partly due to the accumulation of Advanced Glycation Endproducts (AGEs) and the stiffening of the myocardium and arteries. New medication has been developed to break these AGE-crosslinks to improve cardiovascular compliance. The positive influence of regular physical activity is well known for cardiovascular disease and aging. Therefore, what is the most effective intervention, physical exercise and/or new medication AGE-crosslink breakers, in improving the cardiovascular and cerebrovascular compliance and improving the endothelial function in healthy sedentary elderly.

ELIGIBILITY:
Inclusion Criteria:

* Healthy sedentary elderly
* Age 65 yrs and older

Exclusion Criteria:

* Cardiovascular disease
* Cerebrovascular disease
* Changes on ECG indicating cardiomyopathy or ischemia
* No cardiovascular medication
* Diabetes Mellitus
* Hypercholesterolemia
* BMI > 33 kg/m2
* Intensive exercise > 1 hour a week

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Examine the combined effects of one year exercise training and the AGE-crosslink breaker Alagebrium on vascular endothelial function. | 0 and 12 months
  At baseline and 12 months the endothelial function will be measured with an invasive vascular function measurement using the leg model. Via an arterial line in the common femoral artery acethylcholine, sodium nitroprusside and LNMMA will be infused at different dosages. Vascular response will be measured using venous occlusion plethysmography. Non-invasive vascular measurements, e.g.flow mediated dilation and pulse wave velocity, using ultrasound techniques will be performed at 0, 6 and 12 months. Also, cardiopulmonary fitness level will be tested at 0, 3, 6 and 12 months with an ergometer.

SECONDARY OUTCOMES:
Examine the individual effects of one year exercise training and the AGE-crosslink breaker Alagebrium on vascular endothelial function. | 0 and 12 months
  At baseline and 12 months the endothelial function will be measured with an invasive vascular function measurement using the leg model. Via an arterial line in the common femoral artery acethylcholine, sodium nitroprusside and LNMMA will be infused at different dosages. Vascular response will be measured using venous occlusion plethysmography. Non-invasive vascular measurements, e.g.flow mediated dilation and pulse wave velocity, using ultrasound techniques will be performed at 0, 6 and 12 months. Also, cardiopulmonary fitness level will be tested at 0, 3, 6 and 12 months with an ergometer.
Examine the combined effects of one year exercise training and the AGE-crosslink breaker Alagebrium on cardiac function. | 0, 6 and 12 months
  An echocardiogram will be performed at baseline, 6 and 12 months. Measures such as strain, strain rate and myocardial velocity, together with the diastolic function parameters (e.g. E/A, S/D, and E/E' ratio) will be specifically evaluated. Also, the common measures such as wall thickness, volumes, etc, will be examined.
Examine the individual effects of one year exercise training and the AGE-crosslink breaker Alagebrium on cardiac function. | 0, 6 and 12 months
  An echocardiogram will be performed at baseline, 6 and 12 months. Measures such as strain, strain rate and myocardial velocity, together with the diastolic function parameters (e.g. E/A, S/D, and E/E' ratio) will be specifically evaluated. Also, the common measures such as wall thickness, volumes, etc, will be examined.
Examine the combined effects of one year exercise training and the AGE-crosslink breaker Alagebrium on cerebral perfusion and cognitive function. | 0 and 12 months
  A cerebral perfusion measurement will be performed at baseline and after 12 months with transcranial doppler, near infra-red spectroscopy and continuous beat to beat blood pressure monitoring using the Finameter during different posture maneuvers and hypo- and hypercapnia. Dynamic cerebral autoregulation and vasoreactivity will be examined.
  Cognitive function will be measured at baseline, 6 and 12 months using the CANTAB.
Examine the individual effects of one year exercise training and the AGE-crosslink breaker Alagebrium on cerebral perfusion and cognitive function. | 0 and 12 months
  A cerebral perfusion measurement will be performed at baseline and after 12 months with transcranial doppler, near infra-red spectroscopy and continuous beat to beat blood pressure monitoring using the Finameter during different posture maneuvers and hypo- and hypercapnia. Dynamic cerebral autoregulation and vasoreactivity will be examined.
  Cognitive function will be measured at baseline, 6 and 12 months using the CANTAB.

CONTACTS AND LOCATIONS:
Overall Officials: Maria TE Hopman, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Derived] Oudegeest-Sander MH, Olde Rikkert MG, Smits P, Thijssen DH, van Dijk AP, Levine BD, Hopman MT. The effect of an advanced glycation end-product crosslink breaker and exercise training on vascular function in older individuals: a randomized factorial design trial. Exp Gerontol. 2013 Dec;48(12):1509-17. doi: 10.1016/j.exger.2013.10.009. PMID 24400341